CLINICAL TRIAL: NCT05866224
Title: Effects of a Telerehabilitation Program and Detraining on Cardiorespiratory Fitness in Patients With Post-COVID-19 Sequelae
Brief Title: Telerehabilitation Program and Detraining in Patients With Post-COVID-19 Sequelae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus docent Sant Joan de Déu-Universitat de Barcelona (Other)
Responsible Party: Principal Investigator, Manuel Vicente Garnacho Castano, Coordinator of the DAFNiS research group, Campus docent Sant Joan de Déu-Universitat de Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Hospital of Mataró
Record Dates: First submitted 2023-05-16; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised home telerehabilitation program (Experimental): COVID-19 patients will perform a total of 15 weeks of a telerehabilitation program combined with aerobic and strength exercises using the circuit training methodology. COVID-19 patients will carry out 3 weekly sessions on non-consecutive days to avoid unnecessary overload and maximize the adaptations, completing a total of 45 sessions
  Interventions: Other: Telerehabilitation program
- non-supervised control group (No Intervention): COVID-19 patients that will not perform the telerehabilitation program

INTERVENTIONS:
Other: Telerehabilitation program — The supervised telerehabilitation program will be performed in the home of each patient and supervised by an experienced physiotherapist with more than 4 years of clinical experience in therapeutic exercise for chronic diseases.
  Arms: Supervised home telerehabilitation program

SUMMARY:
The primary objective of this study is to evaluate the effects of a 15-week home telerehabilitation program and a detraining period on cardiorespiratory fitness and muscular efficiency in patients with post-COVID-19 sequelae compared to a control group of COVID-19 patients. We hypothesize that cardiorespiratory fitness and muscular efficiency significantly improve in patients who carry out the home telerehabilitation program. However, the cardiorespiratory and muscular adaptations achieved and tolerance to exercise are lost over time as an effect of detraining.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* molecular diagnosis (reverse transcription polymerase chain reaction [RT-PCR]) of infection by SARS-CoV-2
* post-COVID-19 symptomatology

Exclusion Criteria:

* severe neurological disease
* active oncological disease
* neuromuscular disease and/or orthopedic disorders impeding normal development of cardiopulmonary exercise test
* the absence of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness: absolute oxygen uptake | 1 week per group
  absolute peak oxygen uptake in L/min
Cardiorespiratory fitness: relative oxygen uptake | 1 week per group
  relative peak oxygen uptake in L/min
Exercise capacity during cardiopulmonary exercise test | 1 week per group
  Exercise time in minutes and seconds
Mechanical efficiency | 1 week per group
  Delta efficiency in percentage
Ventilatory efficiency | 1 week per group
  VE/VCO2 slope
Power output during pedaling | 1 week per group
  Power output in watts

SECONDARY OUTCOMES:
Respiratory exchange ratio | 1 week per group
  RER
Minute ventilation | 1 week per group
  Ventilation in L/min
ventilatory equivalent for oxygen | 1 week per group
  VE/VO2
ventilatory equivalent for carbon dioxide | 1 week per group
  VE/VCO2
End-tidal partial pressure of oxygen | 1 week per group
  PetO2 in mmHg
end-tidal partial pressure of carbon dioxide | 1 week per group
  PetCO2 in mmHg
Weight of COVID-19 patients | 1 week per group
  Weight in kg
Height of COVID-19 patients | 1 week per group
  Height in meters
Body mass index of COVID-19 patients | 1 week per group
  BMI in kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- Manuel Vicente Garnacho Castaño, Sant Boi de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet decided